CLINICAL TRIAL: NCT07280988
Title: The Effect of Environment Specific Slip Resistant Footwear - A Randomized Cross-Over Study From Danish Dairy Industry
Brief Title: Effectiveness of Slip Resistant Footwear in Dairy Industry
Acronym: SRFDI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Herning Hospital (Other); Sika footwear (Unknown); billigarbejdstøoj.dk (Unknown); Arla Foods (Industry)
Responsible Party: Principal Investigator, Lasse Jakobsen, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20235100802
Record Dates: First submitted 2025-08-29; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Slips; Falls Prevention; Perceived Slipperiness
Keywords: occupational slips; sllips trips and falls; footwear; friction; ergonomics

STUDY DESIGN:
Intervention Model Description: All participants will complete two test sessions: 1) 10 working days in one pair of safety shoes followed by 2) 10 working days in another pair of safety shoes.
  Participants are randomized to start with one pair or the other. Participants will be instructed to resume their normal working routine throughout the study period. All participants will fill out questionnaires every day for the 20 days of testing
Who Masked: Participant
Masking Description: Participants are not made aware of which shoe pair range the best in the laboratory studies. However, no masking of the shoes visual appearance are made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sika shoe (Experimental)
  Interventions: Device: Environment specific safety footwear
- Airtox shoe (Active Comparator)
  Interventions: Device: Environment specific safety footwear

INTERVENTIONS:
Device: Environment specific safety footwear — The participants will wear two different safety shoes (SIKA Highline and AIRTOX FW44) in the test periode (20 working days). 10 working days in each safety shoes.

SUMMARY:
In the dairy industry, same-level falls are a major problem and a well-known challenge. At Arla's dairy in Taulov, where this RCT study is being carried out, reports of risk observations, near incidents, and workplace accidents have increased over the past five years. Accident statistics further show that same-level falls are the most common incidents, with slippery floors and surfaces being by far the main cause of both near incidents and risk observations. Because of this, it is necessary to test different types of safety footwear that, based on laboratory studies, are considered particularly suitable for the working environment in a dairy.

it is hypothesized that employees, through subjective questionnaires, will rate one shoe as less slippery than the other. At the same time, it is hypothesized that employees will also subjectively find one shoe more comfortable than the other.

DETAILED DESCRIPTION:
Slipping, tripping, and falling (STF) are the second most common risk factor for serious occupational accidents in Denmark, accounting for 18.9% of the cases. In fact, general fall accidents in 2016 were estimated to cause annual additional costs of 3.9 billion DKK due to lost productivity, and a further 4.8 billion DKK in healthcare and long-term care expenses. Similar numbers are observed in the United States, where STF is likewise reported as the second most common cause of workplace accidents. The primary cause of STF incidents is often insufficient friction between footwear and walking surfaces. In response to this issue, ASTM International in 2021 raised the minimum threshold for certified slip-resistant footwear, making it even more challenging for manufacturers to meet test requirements. Although recent years have brought advances in the understanding of mechanisms leading to STF events-particularly slipping-there is still insufficient research translating this knowledge into practical preventive measures. Data from the Danish Working Environment Authority confirm this gap, showing that reported STF accidents increased between 2016 and 2021. Moreover, the actual number of near incidents is likely even higher, as many are never formally registered. Implementing existing prevention knowledge into effective, practical interventions remains a key challenge. Analysis of gait patterns has been suggested as a way to better understand changes in walking stability, thereby enabling quantification of near-incidents occurrences.

This RCT study will, for the first time, combine multiple measurement parameters, including reported falls, near incidents, risk situations, perceived slip resistance, and gait characteristics (e.g., step length, cadence). These outcomes will be measured through both quantitative and qualitative methods. Quantitative gait data will be collected using accelerometers, with two sensors allocated to each participants foot/shoe. This system has previously been used to quantify gait patterns. Qualitative data will be collected through self-reported records. By linking spatiotemporal gait parameters with self-reported accident and near-miss data, this study will provide new insights into the relationship between objective and subjective safety outcomes. In addition, it is crucial to identify potential barriers and challenges experienced both by employees using slip-resistant footwear and by procurement decision-makers responsible for footwear acquisition. To address this, focus group interviews and surveys will be conducted among study participants as well as procurement staff at Arla in Taulov.

A power calculation estimated the required sample size at 28 participants, based on an expected α of 0.05, β of 0.20, and an effect size of 0.25. Allowing for an anticipated dropout rate of 20%, the recruitment target is set at 34 participants (17 in each study arm). Considering the number of employees working in slippery zones, it was decided that only a cross-over design will enable to recruit a sufficient number of participants. Employees at Arla's Taulov dairy will be recruited and randomized (1:1) to either start working with one pair of safety shoes while the other half will start with the other pair of safety shoes using a computer-generated minimization sequence, ensuring balance between groups in terms of sex, age, and prior fall history.

Quantitative and qualitative data will be presented descriptively. Following a thematic analysis approach, outcomes such as comfort, gait patterns, perceived safety, fall/near-fall experiences, and economic considerations (e.g., purchase costs) will be displayed in a structured format that provides an overview of participants' experiences of the intervention as well as perceived barriers and benefits. To evaluate changes over time, quantitative outcomes will be analyzed using two-way repeated measures ANOVA. Multiple imputation will be used to handle potential missing data, and differences between groups will be further assessed using post-hoc tests.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employed at Arla Taulov dairy facility.
* No major injuries affecting their daily work.
* No plans of retiring before the end of the study period.

Exclusion Criteria:

* Surgery in the feet and under extremity within the last three months. Pregnancy.
* Part-time workers.
* Neurological disorders affecting gait.
* Can read and understand Danish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Self-reported feel of slipperines | Through study completion, an average of 20 working days
  Self-rated feel of slipperiness. "To what extent did you feel the need to walk carefully today?" Rated on a continuous VAS scale (not slippey to the right and slippery to the left). Less slippery towards right and most slippery towards left. Hence, towards right is better. These are obtained with daily questionaries.

SECONDARY OUTCOMES:
Spatiotemporal gait characteristics | Through study completion, an average of 20 working days
  Step length will be obtained using accelerometers positioned on the participants' shoes. This will be measured in meters.
Slipping without falling | Through study completion, an average of 20 working days
  "Did you experience a slip today without falling?" These are obtained with daily questionaries. Yes/No
Slipping and falling | Through study completion, an average of 20 working days
  "Did you experience a slip today resulting in a fall?" These are obtained with daily questionaries. Yes/No

OTHER OUTCOMES:
Working hours | through study completion, an average of 20 working days
  "How many hours did you work today?" These are obtained with daily questionaries.
Division of work | Through study completion, an average of 20 working days.
  "In which division did you work today?" Choose between kit warehouse, packing, cheese factory or process. These are obtained with daily questionaries.
Floor type | Through study completion, an average of 20 working days.
  "How much of your workday today did you spend on dry floors, wet floors and greasy floors?" Reported in hours. These are obtained with daily questionaries.
Comfort | After 10 working days.
  "Overall, how comfortable have you found the shoes you have worn over the past 10 workdays?" Rated on a continuous visual analog scale (comfort to the right and discomfort to the left). These are obtained with questionaries after wearing one shoe for 10 working days.
General slipperiness | After 20 working days.
  "Overall, how have you experienced the slip resistance of the shoes you have worn during the past 10 workdays?" These are obtained with questionaries after wearing one shoe for 10 working days. Rated on a continuous visual analog scale (not slippey to the right and slippery to the left).

CONTACTS AND LOCATIONS:
Locations (1):
- Arla Foods AMBA, Taulov, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redfern MS, Cham R, Gielo-Perczak K, Gronqvist R, Hirvonen M, Lanshammar H, Marpet M, Pai CY, Powers C. Biomechanics of slips. Ergonomics. 2001 Oct 20;44(13):1138-66. doi: 10.1080/00140130110085547. PMID 11794762
- [Background] Chang WR, Gronqvist R, Leclercq S, Myung R, Makkonen L, Strandberg L, Brungraber RJ, Mattke U, Thorpe SC. The role of friction in the measurement of slipperiness, Part 1: friction mechanisms and definition of test conditions. Ergonomics. 2001 Oct 20;44(13):1217-32. doi: 10.1080/00140130110085574. PMID 11794765
- [Background] ASTM International, "Standard Specification for Performance Requirements when Evaluating Slip Resistance of Protective (Safety) Footwear using ASTM F2913 Whole Shoe Test Method.
- [Background] L. Strandberg and H. Lanshammar, "The dynamics of slipping accidents," J. Occup. Accid., vol. 3, pp. 153-162, 1981,
- [Background] Hanson JP, Redfern MS, Mazumdar M. Predicting slips and falls considering required and available friction. Ergonomics. 1999 Dec;42(12):1619-33. doi: 10.1080/001401399184712. PMID 10643404
- [Background] Gronqvist R, Chang WR, Courtney TK, Leamon TB, Redfern MS, Strandberg L. Measurement of slipperiness: fundamental concepts and definitions. Ergonomics. 2001 Oct 20;44(13):1102-17. doi: 10.1080/00140130110085529. PMID 11794760
- [Background] GBD 2021 Causes of Death Collaborators. Global burden of 288 causes of death and life expectancy decomposition in 204 countries and territories and 811 subnational locations, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2024 May 18;403(10440):2100-2132. doi: 10.1016/S0140-6736(24)00367-2. Epub 2024 Apr 3. PMID 38582094
- [Background] Sundhedsstyrelsen, "Sygdomsbyrden i Danmark, Ulykker, Selvskade og Selvmord 2016," Copenhagen S, 2016.
- [Background] Beskæftigelsesministeriet, "Et nyt og forbedret arbejdsmiljø - Bilagsrapport, Bind 1," 2018.